CLINICAL TRIAL: NCT05658484
Title: A Multicenter, Postmarketing Study of Dimethyl Fumarate (Tecfidera; BG00012) in Relapsing Forms of Multiple Sclerosis (RMS) Participants in China
Brief Title: A Study of Dimethyl Fumarate (DMF) in Relapsing Forms of Multiple Sclerosis (RMS) Participants in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109MS424
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dimethyl fumarate (DMF) (Experimental): Participants will receive DMF 120 mg capsules, orally, twice daily (BID) for the first 7 days, followed by 240 mg BID (maintenance dose) after 7 days for up to Week 48.
  Interventions: Drug: Dimethyl fumarate

INTERVENTIONS:
Drug: Dimethyl fumarate — Administered as specified in the treatment arm.
  Other Names: Tecfidera; DMF; BG00012

SUMMARY:
The primary objective of the study is to assess the efficacy of DMF in Chinese participants with RMS at Week 48. The secondary objectives of the study are to assess the efficacy and safety of DMF in Chinese participants with RMS.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a baseline (pre-dose on Day 1) Expanded Disability Status Scale (EDSS) between 0.0 and 5.0, inclusive.
* Must have experienced at least 1 documented relapse within the 12 months before screening, with a prior brain magnetic resonance imaging (MRI) demonstrating lesion(s) consistent with MS or have showed evidence of GdE lesion(s) of the brain on an MRI performed within the 6 weeks prior to screening.

Key Exclusion Criteria:

* An MS relapse that occurred within the 30 days prior to screening and/or the participant has not stabilized from a previous relapse prior to screening.
* Current hepatitis C infection and current hepatitis B infection. Participants with immunity to hepatitis B from previous natural infection or vaccination are eligible to participate in the study.
* History of severe allergic or anaphylactic reactions or of any allergic reactions that, in the opinion of the Investigator, are likely to be exacerbated by any component of the study treatment.
* History or positive test result at screening for human immunodeficiency virus (HIV).
* Use at the time of enrollment and/or anticipated ongoing use of any traditional and/or unlicensed medicines and/or traditional therapies and/or herbal preparations, which are known or considered by the Investigator to affect MS and endpoints that are being considered in the study, including safety and efficacy.
* Current enrollment in any other investigational drug study or participation in any other investigational study within 6 months prior to screening.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-04-12 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | Week 48
  ARR is defined as the number of confirmed MS relapses in a year. MS relapse is defined as new or recurrent neurologic symptoms, not associated with fever or infection, lasting for at least 24 hours, accompanied by one or more of the following: New objective neurological findings upon examination by the treating neurologist that are functionally consistent with findings on the Expanded Disability Status Scale (EDSS) (performed within 5 days of onset of symptoms) with an increase over the prior visit of ≥0.5 for the total score, an increase of ≥2 in 1 functional system (FS), except bladder/cognitive changes, and/or an increase of ≥1 in 2 FS, except bladder/cognitive changes

SECONDARY OUTCOMES:
Change From Baseline in Number of Gadolinium-Enhancing (GdE) Lesions | Week 24
Number of GdE Lesions | Week 24 and 48
Percentage of Participants GdE-Lesion Free | Week 24 and 48
Percentage of Participants Relapsed | Week 48
Number of New T1 Hypo-Intense Lesions | Baseline, Week 24 and 48
Number of New/Newly Enlarging T2 Hyperintense Lesions | Baseline, Week 24 and 48
Total T2 Lesion Volume | Week 24 and 48
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 50
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, in the view of the Investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect and is a medically important event.
Number of Participants With Change from Baseline in Clinical Laboratory Parameters, Electrocardiogram (ECG), and Vital Signs | Baseline to Week 48
Number of Participants With Columbia-Suicide Severity Rating Scale (C-SSRS) Events | Baseline to Week 48
  The C-SSRS is a clinician-administered instrument that systematically assess suicidal ideation and behavior rating scale. It rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent). The scale identifies specific behaviors ranging from "preparatory acts or behavior" to "suicide" which may be indicative of an individual's intent to complete suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (15):
- China (15):
  - Beijing Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - The Second Hospital of Hebei Medical University, Hebei
  - The First People's Hospital of Yunnan Province, Kunming
  - Renji Hospital, Shanghai Jiatong Uni. School of Medicine, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - The First Hospital of China Medical University, Shengyang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Second Affiliated Hospital of Air Force Medical University, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/